CLINICAL TRIAL: NCT07150819
Title: Effectiveness of a Multidisciplinary Perioperative Pain Management Model in Enhancing Recovery After Anorectal Surgery
Brief Title: A Multidisciplinary Perioperative Pain Management
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This research plan needs to be readjusted.
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Ying Zhang, Associate Chief Physician, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ChinaJapanFH010
Record Dates: First submitted 2025-08-28; First posted 2025-09-02 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Anorectal Surgery; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Standard Nursing Care
  Interventions: Behavioral: Standard Nursing Care Protocol
- Observation Group (Experimental): MDC-based Pain Management
  Interventions: Behavioral: MDC-based Pain Management

INTERVENTIONS:
Behavioral: Standard Nursing Care Protocol — The control group received standard perioperative nursing care in accordance with the Chinese Consensus and Clinical Guidelines for Enhanced Recovery After Surgery (2021 edition) and the Expert Consensus on Perioperative Nursing of Anorectal Diseases (2022 edition). Preoperative fasting included a 6-hour restriction on solid food and a 2-hour restriction on clear liquids. At 8:00 p.m. on the night before surgery, patients were instructed to orally ingest 500 mL of 10% glucose solution to supplement energy reserves. Fifteen minutes of structured health education was delivered preoperatively by the assigned nurse using 3D animations to explain the surgical process. Intraoperatively, an inflatable warming blanket was used to maintain the core temperature at 38°C, and all infusion fluids were pre-warmed to 37°C. For infection prophylaxis, 30 minutes before incision, patients received intravenous cefazolin (1 g for body mass index [BMI] < 25 kg/m²; 2 g for BMI ≥ 25 kg/m²).
  Arms: Control Group
Behavioral: MDC-based Pain Management — In accordance with the IASP Guidelines for Multidisciplinary Postoperative Pain Management (2023) and the Expert Consensus on Multidisciplinary Collaboration for Pain Management in China, a three-tier MDC framework was established;Surgeons were responsible for optimizing surgical procedures (e.g., using the tissue selecting technique for stapled hemorrhoidectomy) and administering a local injection of 5 mL 0.25% ropivacaine around the wound margin at the end of surgery. Anesthesiologists performed preoperative ASA physical status classification, monitored intraoperative vital signs, and configured postoperative patient-controlled analgesia (PCA) with sufentanil at 0.02 μg/kg/h.Compound Methylene Blue Nerve Block: A solution was prepared by mixing 2 mL of 1% methylene blue, 10 mL of 0.75% ropivacaine, and 8 mL of normal saline, yielding final concentrations of 0.02% methylene blue and 0.25% ropivacaine.
  Arms: Observation Group

SUMMARY:
Objective: This study aimed to evaluate the clinical value of a multidisciplinary collaboration (MDC)-based perioperative pain management model. Methods: A prospective, randomized controlled trial was conducted involving 126 patients who underwent anorectal surgery between July 2022 and December 2023. Participants were randomly assigned (1:1) using a computer-generated sequence to either the control group (n = 63), which received standard nursing care, or the observation group (n = 63), which received nursing care based on the MDC model integrating surgery, anesthesiology, nursing, psychology, and pharmacy disciplines.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years (adult patients capable of cooperating with assessments and interventions; pediatric patients were excluded due to developmental differences in pain perception and response);
* No severe anal malformations (defined as conditions that could significantly alter surgical technique or affect wound healing, such as anal stenosis or grade III or higher rectal prolapse) and no history of previous anal surgery;
* Complete clinical data available;
* Clear consciousness and intact cognitive and communication abilities, with the capacity to comply with study assessments and interventions;
* Diagnosis of a common benign anorectal disease requiring elective surgery (e.g., grade III/IV mixed hemorrhoids, simple anal fistula, chronic anal fissure, low perianal abscess) in accordance with the diagnostic criteria outlined in the Guideline for Clinical Diagnosis and Treatment of Hemorrhoids (2017 edition).

Exclusion Criteria:

* Diagnosis of inflammatory bowel disease, colorectal malignancy, or active intestinal infection; presence of significant dysfunction in major organs (e.g., ASA [American Society of Anesthesiologists] physical status classification ≥ III), autoimmune diseases, or long-term use of immunosuppressants or corticosteroids;
* History of chronic pain syndromes or long-term use of opioid analgesics;
* Presence of moderate-to-severe lumbar spinal disease or deformity that precludes neuraxial anesthesia (e.g., planned spinal anesthesia);
* Withdrawal from the study or incomplete clinical data;
* History of psychiatric disorders or cognitive impairment rendering the patient unable to comply with assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Short-Form McGill Pain Questionnaire (SF-MPQ) | 4 hours
  The SF-MPQ includes two core components: the pain rating index (PRI) and present pain intensity (PPI). The PRI assesses the qualitative aspects of pain using 11 sensory descriptors (e.g., stabbing, throbbing) and 4 affective descriptors (e.g., fearful, exhausting), with a total score ranging from 0 to 45. The PPI is a single-item, 6-point scale (0 = no pain, 5 = excruciating pain).
Dynamic Pain Intensity Monitoring | 4 hours
  The VAS [27] was used to assess pain intensity at five postoperative time points: immediately after surgery (T0), and at 4 hours (T1), 12 hours (T2), 24 hours (T3), and 48 hours (T4) postoperatively. The VAS consists of a 10 cm horizontal line anchored by "no pain" at 0 cm and "worst possible pain" at 10 cm; patients were asked to mark the point that best reflected their current pain level. The mark was then converted into a numeric score ranging from 0 to 10. Pain intensity was categorized as follows: 1-3 (mild, does not interfere with daily activities), 4-6 (moderate, interferes with sleep), and 7-10 (severe, completely disabling). The scale demonstrated strong internal consistency (ICC = 0.89, P < 0.001) and high concurrent validity with the Numerical Rating Scale (r = 0.94)
Postoperative Recovery Indicators | 4 hours
  Four objective time-based recovery parameters were recorded: (1) Time to first defecation, defined as the number of hours from anesthesia recovery to the first spontaneous bowel movement; (2) Time to first ambulation, defined as the time postoperatively at which the patient could independently stand and walk for ≥5 minutes; (3) Wound healing time, defined as the number of days required for complete epithelialization and absence of exudate, as confirmed by blinded assessment by the attending physician; (4) Length of postoperative hospital stay, measured in calendar days from the end of surgery to the date of discharge documentation.
Postoperative Complication Monitoring | 1 Day
  Postoperative complications within 30 days were identified and recorded based on internationally accepted diagnostic criteria: (1) Urinary retention, defined as a bladder volume >400 mL on ultrasound requiring catheterization (per the International Continence Society standard); (2) Perianal edema, defined as a palpable perianal bulge ≥1 cm in diameter with tenderness, confirmed via blinded physician assessment; (3) Wound infection, meeting criteria established by the Centers for Disease Control and Prevention (erythema, swelling, warmth, pain, and purulent discharge or white blood cell count >10×10⁹/L); (4) Constipation, defined as no defecation within 72 hours postoperatively requiring pharmacological intervention (Rome IV criteria); (5) Anal distension, characterized by persistent anal pressure or fullness with a VAS score ≥4 sustained for more than 24 hours.
Psychological Status Assessment | 1 day
  The DASS-21 [30] was used to evaluate psychological well-being, comprising three subscales: depression (7 items), anxiety (7 items), and stress (7 items). Each item is rated on a 4-point Likert scale from 0 ("Did not apply to me at all") to 3 ("Applied to me very much or most of the time"). Assessments were conducted at two time points: 24 hours preoperatively (baseline) and on day 7 postoperative (post-intervention). The Chinese version of the DASS-21 has demonstrated high internal consistency in postoperative patient populations: Cronbach's α = 0.89 for depression, α = 0.84 for anxiety, and α = 0.87 for stress. Confirmatory factor analysis supported good model fit (comparative fit index = 0.92, root mean square error of approximation = 0.06)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhang, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospita, Beijing, Beijing City, China

IPD SHARING:
Plan to Share IPD: No